CLINICAL TRIAL: NCT06752226
Title: Effect of Action Observation Training on Gross Motor Function in Children with Spastic Cerebral Palsy
Brief Title: Effect of AO Training on Gross Motor Function in Children with Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ekram magdy Mohamed fadl, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: exercises on motor function
Record Dates: First submitted 2024-12-21; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Diplegic Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic

STUDY DESIGN:
Intervention Model Description: parallel study is a type of clinical study in which two or more groups of participations receive different interventions
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Effect of action observation training on gross motor function in children with cerebral palsy (Experimental): Action observation training used to improve gross motor function including walking, jumping and running domain in children with cerebral palsy by observing at imitate phases of gait cycle performed by a normal person
  Interventions: Other: action observation trainingAOT refers to an observational practice that has been used extensively for the goal of motor programming and enhances motor learning and performance
- action observation training (Experimental): Action observation training (AO) is cognitive intervention technique that is used to improve and learn exercise skills in sports, athletes, the general public and patient with motor impairment
  Interventions: Other: action observation trainingAOT refers to an observational practice that has been used extensively for the goal of motor programming and enhances motor learning and performance

INTERVENTIONS:
Other: action observation trainingAOT refers to an observational practice that has been used extensively for the goal of motor programming and enhances motor learning and performance — In AOT, motor-related information can be available through the visual function by encoding into the mental representation of the memory to organize the intended action

SUMMARY:
The study was conducted to examine the impact of the action observation training (AOT) on gross motor function in children with spastic cerebral palsy.

DETAILED DESCRIPTION:
Thirty children with spastic diplegic cerebral palsy aged from 4 to 7 years were randomly allocated into two groups of equal number; study group (A) and control group (B). Both groups received designed physical therapy program for 45 minutes, three times/ per week for two successive months. In addition, study group received action observation (AO) training for 30 minutes per session. All phases of gait cycle and functional ability of all children participating in both groups was assessed by kenovia software and gross motor function measure (GMFM) walking, running and jumping domain.

ELIGIBILITY:
Inclusion Criteria:

Age ranges from 4 - 7 years. Level Ι - Π according to Gross Motor Functional Classification System (GMFCS) (Appendix II).

Grade 1, +1 and 2 of the Modified Ashworth Scale (Appendix III). Able to follow verbal commands and instructions.

Exclusion Criteria:

* Significant visual or auditory impairments Structural or fixed soft tissue deformities of Lower extremities. Perception disorders. Botox injection in the lower extremity in the past 6 months.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-05-27 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 8 weeks
  1. Gross Motor Function Measure All children were assessed using the GMFM-88 scale. The GMFM scale has been validated to assess change in motor performance in children with CP. In this study we assessed the items of walking, running and jumping of the GMFM. The items are scored on four-point ordinal scales (0=cannot initiate; 1=initiates; 2=partially completes item; 3=completes item independently)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy , Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided